CLINICAL TRIAL: NCT06713200
Title: Effectiveness Of The Application Of Percutaneous Electrolysis On Muscular Scar Tissue Of The Medial Gastrocnemius: A Doble-Blinded Randomized Clinical Trial
Brief Title: Effectiveness Of The Application Of Percutaneous Electrolysis On Muscular Scar Tissue.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Carlos Vicente Vega, Graduated in physiotherapy, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI 2023 08 1418 - TD
Record Dates: First submitted 2024-11-20; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Muscle Injury; Fibrosis
Keywords: TENNIS LEG; GASTROCNEMIOUS INJURY; FIBROSIS; PERCUTANEOUS ELECTROLYSIS
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Intervention Model Description: The study will include pacients randomized into three treatment groups: high-intensity percutaneous electrolysis, low-intensity and a control group with sham treatment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects treated with high-intensity percutaneous electrolysis. (Active Comparator)
  Interventions: Procedure: High intensity percutaneous electrolysis
- Subjects treated with low intensity percutaneous electrolysis. (Active Comparator)
  Interventions: Procedure: Low intensity Percutaneous Electrolysis
- Subjects treated with simulated percutaneous electrolysis (Sham Comparator)
  Interventions: Procedure: Simulated Percutaneous Electrolysis

INTERVENTIONS:
Procedure: High intensity percutaneous electrolysis — A sterile, disposable stainless steel needle of different lengths depending on the area to be treated will be connected to the EP device; the gauge of these needles will be 0.25 mm. A current of 3 mA will be applied for 3 times with a duration of 3 seconds each. In order to avoid biases, the technique will be performed for 90 seconds as in the low intensity treatment group and in the last 20 seconds the current will be applied with the parameters previously described. Three sessions divided in three consecutive weeks will be applied.
  Arms: Subjects treated with high-intensity percutaneous electrolysis.
Procedure: Low intensity Percutaneous Electrolysis — This technique will be performed with the same instrument as the high intensity technique. It differs from the previous treatment group in that the current intensity in this case will be of an amperage of 0.3mA during 90 seconds. In the same way, 3 sessions divided in 21 consecutive days will be applied.
  Arms: Subjects treated with low intensity percutaneous electrolysis.
Procedure: Simulated Percutaneous Electrolysis — The needle and PD device will be connected in the same way as for the other treatment groups. The needle will be inserted without reaching the lesion area and the characteristic sound of turning on the PD machine will be made. It will last 90 seconds and at no time the galvanic current will be applied. The same aseptic precautions will be applied, in addition to performing the same final hemostasis guidelines and providing the same post-treatment guidelines as for all the other subjects in the study.
  Arms: Subjects treated with simulated percutaneous electrolysis

SUMMARY:
OBJECTIVE: Determine the effectiveness of an intervention that consists of the application of percutaneous electrolysis in different doses compared to the application of a simulated intervention in adults who present a muscle tear in the internal gastrocnemius.

MATERIAL AND METHODS: Around fifty adults with muscle tears in the medial gastrocnemius will be included in the following study. The first group will be treated with high-intensity percutaneous electrolysis (3 mA), the second group will be treated with low-intensity percutaneous electrolysis (0.3 mA), and the third group will receive a sham intervention. Myofascial pain, level of kinesiophobia, range of ankle dorsiflexion with full knee extension, and triceps surae muscle fatigue will be evaluated both before and after treatment.

APPLICABILITY OF THE EXPECTED RESULTS: The results of this study are intended to help provide information about the effects of electrolysis on muscle tears, thus improving their management. Likewise, this work can contribute to the knowledge of the use of percutaneous electrolysis since it applies two protocols with different intensity and application time. In this way, it will provide information on the treatment, management and prognosis of muscle injuries addressed through invasive physiotherapy and more specifically, percutaneous electrolysis.

ELIGIBILITY:
Inclusion Criteria:

* Muscle injury in the medial gastrocnemius
* Pain in the area of injury
* Informed of the purpose, risks and benefits of this study and written consent to participate in the trial.

  * Available for follow-up.

Exclusion criteria:

* Active rehabilitation for another musculoskeletal pathology.
* Belenophobia
* Immunosuppression.
* Uncontrolled metabolic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Pain at rest | From admission to the end of treatment at 28 days
  Pain assessment of participants' pain in both upright and contracted positions will be performed using a 10-point Verbal Numerical Pain Scale (0=no pain, 10=maximum pain tolerable). Subjects will be asked to rate numerically the pain at rest and in a maintained position of elevation of both heels, also commonly known as "standing on tiptoe". In the latter position, 10 will be considered if the subjects fail to stand in this position for at least one complete elevation.
Pain on load | From admission to the end of treatment at 28 days
  Pain assessment of participants' pain in both upright and contracted positions will be performed using a 10-point Verbal Numerical Pain Scale (0=no pain, 10=maximum pain tolerable). Subjects will be asked to rate numerically the pain at rest and in a maintained position of elevation of both heels, also commonly known as "standing on tiptoe". In the latter position, 10 will be considered if the subjects fail to stand in this position for at least one complete elevation.
Level of kinesiophobia | From admission to the end of treatment at 28 days
  Recovery from painful injuries is associated with fear of movement or also called kinesiophobia. It could be defined as an irrational or excessive fear of movement for fear of injury or re-injury. That is why a kinesiophobia questionnaire (Annex II) will be provided at the beginning of the study (day I, assessment and first intervention) to all participants to assess kinesiophobia to perform certain movements that may cause pain or worsen previous injuries. It consists of 11 questions with a minimum score of 11 and a maximum score of 44.
Ankle dorsiflexion range with the knee in extension. | From admission to the end of treatment at 28 days
  The evaluation of this variable will be carried out by measuring the angle extracted from the dorsiflexion of the ankle with a knee extension. This stretch is commonly performed in sports practice so patients are generally already familiar with it. The stretches will be performed with the participants barefoot. Likewise, the participants will be instructed on the positioning of the test. The leg to be evaluated will be placed in such a way that the foot is placed in the midline of an area marked on the floor, and the foot of the healthy leg will be placed forward at the distance of one step. The end point of the gastrocnemius stretch will be defined as the point at which the participants feel discomfort without lifting the heel and without pelvic rotation.
Muscle fatigue | From admission to the end of treatment at 28 days
  Fatigue in this muscle group will be assessed by performing a heel-raise test at the beginning and end of the trial for all participants who have completed it. The test consists of placing the patient on one leg and, using a metronome at a speed of 40 beats per minute (Garmin Fénix 5/5S), asking them to raise their heels. If they are unable to raise their heels for 3 consecutive beats, fatigue will be considered. Light support on a wall is allowed to maintain the patient's balance.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Barbero-Iglesias, Doctor, Study Director — University of Salamanca
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De-la-Cruz-Torres B, Romero-Rodriguez B, Romero-Morales C. Ultrasound-Guided Percutaneous Needle Electrolysis Combined With Therapeutic Exercise May Add Benefit in the Management of Soleus Injury in Female Soccer Players: A Pilot Study. J Sport Rehabil. 2022 Nov 21;32(3):265-271. doi: 10.1123/jsr.2022-0021. Print 2023 Mar 1. PMID 36410342
- [Background] Lopez-Martos R, Gonzalez-Perez LM, Ruiz-Canela-Mendez P, Urresti-Lopez FJ, Gutierrez-Perez JL, Infante-Cossio P. Randomized, double-blind study comparing percutaneous electrolysis and dry needling for the management of temporomandibular myofascial pain. Med Oral Patol Oral Cir Bucal. 2018 Jul 1;23(4):e454-e462. doi: 10.4317/medoral.22488. PMID 29924769
- [Background] De-la-Cruz-Torres B, Barrera-Garcia-Martin I, Valera-Garrido F, Minaya-Munoz F, Romero-Morales C. Ultrasound-Guided Percutaneous Needle Electrolysis in Dancers with Chronic Soleus Injury: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2020 Aug 27;2020:4156258. doi: 10.1155/2020/4156258. eCollection 2020. PMID 32908559

DOCUMENTS (2):
  • Study Protocol (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT06713200/Prot_000.pdf
  • Informed Consent Form (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT06713200/ICF_001.pdf